CLINICAL TRIAL: NCT07037095
Title: Correlation Between Gastrocnemius Muscle Strain and Functional Performance in Footballers
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: DPT/Batch-Fall20/1005
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Muscle Strain
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ankle plantar flexion test
  Interventions: Diagnostic Test: Ankle plantar flexion test:

INTERVENTIONS:
Diagnostic Test: Ankle plantar flexion test: — Ankle plantarflexion is valid test used to assess for gastrocnemius muscle strain . Patient is asked to actively plantarflex the foot against resistance while examiner Observe ,this action activates the gastrocnemius muscle .The reliability for ankle plantar flexion is 0.81 to 0.99. If the patient reports pain in the region of gastrocnemius, the test is positive. If there is no pain , weakness or difficulty performing plantarflexion then suggest that test is negative.

SUMMARY:
Footballers are highly prone to lower extremity injuries due to the intense physical demands of the sport, with calf muscle strains, particularly gastrocnemius injuries, being very common. The gastrocnemius muscle plays a critical role in movement, posture, and athletic performance.

DETAILED DESCRIPTION:
This study aims to determine the correlation between the severity of gastrocnemius muscle strain and functional performance among footballers. Participants aged 18-40 years with clinically diagnosed gastrocnemius strains were assessed using the Lower Extremity Functional Scale (LEFS) and Hop Test. Severity was categorized through physical examination techniques like palpation, passive dorsiflexion stretch, and resisted plantarflexion tests. Data analysis will explore the relationship between strain severity and functional outcomes, providing valuable insights into rehabilitation strategies and return to play decisions for injured athletes. This study addresses a research gap by focusing specifically on footballers and correlating strain severity with sport-specific functional performance.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients aged between 18 and 40 years.
* At least six months of football training.
* The study focused on players with gastrocnemius muscle injury injuries diagnosed by physical examination; palpation, Stretch Test (Passive Dorsiflexion Test), Resisted Plantarflexion Test.
* Willing to provide written informed consent and comply with study protocols.

Exclusion Criteria:

* Players with Achilles tendon injuries were excluded from the study.
* History of extrinsic trauma
* soleus or other calf injury not meeting inclusion conditions
* Inability to perform rehabilitation
* No intention to return to full sports act

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Footballers are highly prone to lower extremity injuries due to the intense physical demands of the sport, with calf muscle strains, particularly gastrocnemius injuries, being very common.
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Lower Extremity Functional Scale (LEFS) | 6 Month
  The Lower Extremity Functional Scale (LEFS) is a questionnaire used to assess an individual's functional limitations related to their lower extremities. It contains 20 items, each scored on a scale of 0 to 4, with higher scores indicating better function. The total score ranges from 0 to 80, with 80 representing no functional limitations
Hop tests | 6 Months
  The Hop tests are used to assess lower limb function, particularly after injury, and are scored using the Limb Symmetry Index (LSI) by comparing the injured leg's performance to the uninjured leg. A score of 90% or higher on the LSI is generally considered a satisfactory level of recovery, indicating readiness to return to sports.

CONTACTS AND LOCATIONS:
Locations (1):
- Superior university support club, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No